CLINICAL TRIAL: NCT05238753
Title: Electromagnetic Stimulation of the Phrenic Nerve to Generate Contraction of the Diaphragm in Critically Ill Mechanically Ventilated Patients - a Proof-of-concept Study (STIMIT-II)
Brief Title: Electromagnetic Stimulation of the Phrenic Nerve in Critically Ill Mechanically Ventilated Patients (STIMIT-II)
Acronym: STIMIT-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CE certificate ended and was not renewed
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Stimit AG (Industry)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STIMIT-II
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Muscle Weakness; Critical Illness; Mechanical Ventilation Complication
Keywords: VIDD; ICUAW; Muscle Weakness; Weaning
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Intervention Model Description: 15 patients in control group, 15 patients in interventional group with sequential design in term of daily frequency of non-invasive electromagnetic phrenic nerve stimulation, i.e. starting with 5 patients with 2 stimulation per day, followed by 5 patients with 3 stimulations and 5 patients with 5 stimulations per day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, stimulated (Experimental): Electromagnetic stimulation of the phrenic nerve in critically ill patients.
  Interventions: Device: Non-invasive electromagnetic stimulation
- Control, not stimulated (No Intervention): Control group, no stimulation of the phrenic nerve.

INTERVENTIONS:
Device: Non-invasive electromagnetic stimulation — Non-invasive bilateral electromagnetic stimulation of the phrenic nerve
  Arms: Intervention, stimulated

SUMMARY:
Ventilator-induced diaphragmatic dysfunction is a common issue in critically ill patients. Muscle stimulation has shown to have beneficial effects in muscle groups on the extremities. A non-invasive way to stimulate the diaphragm would be the electromagnetic stimulation but it is currently unclear if that is feasible.

In this proof-of-concept trial the primary aim is to show that it is possible to induce a diaphragmatic contraction in critically ill ICU patients via an external electromagnetic stimulation of the phrenic nerve, leading to an inspiration (i) with a sufficient tidal volume (3-6 ml/kg ideal body weight) and (ii) with verifiable muscular diaphragmatic contraction through ultrasound imaging.

DETAILED DESCRIPTION:
During the time of first spontaneous breathing trial 60% of mechanically ventilated patients present with diaphragmatic weakness or also know as ventilator-induced diaphragmatic dysfunction (VIDD). The damage to the diaphragm in terms of muscle atrophy has been shown as early as 12 hours after initiation of mechanical ventilation. Recently, a correlation between diaphragmatic atrophy and mortality could be established.

Induction of diaphragmatic contractions via stimulation of the phrenic nerve would be a possible method to prevent or treat VIDD. A possible modality would be the non-invasive electromagnetic stimulation but feasibility has not been established.

In this proof-of-concept trial the primary aim is to show that it is possible to induce a diaphragmatic contraction in critically ill ICU patients via an external electromagnetic stimulation of the phrenic nerve, leading to an inspiration (i) with a sufficient tidal volume (3-6 ml/kg ideal body weight) and (ii) with verifiable muscular diaphragmatic contraction through ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years old, hospitalized in ICU
* Mechanical ventilation < 36 h
* Prone to stay ventilated > 72 h

Exclusion Criteria:

* Known neurological condition affecting motor neuron or muscle (e.g. ALS)
* Known paralysis of the phrenic nerve
* Proven or suspected spinal cord injury that contraindicates weight bearing on the spinal cord
* Conditions that limit diaphragm movement (high intra-abdominal pressure, ascites, obesity)
* Not able to read and understand the national language German
* Patients with Implanted cardiac support systems (pacemaker, implanted defibrillator)
* Patients with implanted medical pumps
* Pregnant patients
* Patients with skin lesions, infections or strictures in throat/neck area
* Patients with metallic implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Frequency of non-feasible stimulation, due to organisational or patient-specific reasons. | 10 days
  Percentage of non-feasible stimulation out of the total number of stimulations planned according to the investigation protocol.
Time to find the optimal stimulation point of the N. phrenicus | Study duration (10 days)
  Time between first successful N. phrenicus stimulation and identification of the optimal stimulation locus in seconds
Frequency of sufficient Tidal volume generated by electromagentical stimulation of the phrenic nerve (3-6 ml/kg ideal body weight) | Study duration (10 days)
  Percentage of stimulated breaths above the cut-off Today volume (3-6 ml/kg ideal body weigh) out of the total number of stimulated breaths. Tidal volumes are measured by the mechanical ventilator.

SECONDARY OUTCOMES:
Variance of Tidal volume generated by electromagentical stimulation of the phrenic nerve | Study duration (10 days)
  Measurement of variance among the Tidal volumes stimulated during the experimental therapy intervention; Tidal volumes are measured by the mechanical ventilator.
Correlation between amplitude and duration of sEMG signals during stimulated breathing. | Study duration (10 days)
  sEMG amplitude and duration are measured by a device (sEMG Amplificator) connected to electrodes applied to the patient's chest during electromagnetic phrenic nerve stimulation.
Transpulmonary pressure during electromagnetical stimulation of the phrenic nerve | Study duration (10 days)
  Transpulmonary pressure is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Occlusion pressure during electromagnetical stimulation of the phrenic nerve | Study duration (10 days)
  Occlusion pressure is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Diaphragm thickening fraction | approx. 28 days (till ICU discharge)
  Diaphragm thickening fraction measured with ultrasound of the diaphragm.
Diaphragm excursion | approx. 28 days (till ICU discharge)
  Diaphragm excursion measured with ultrasound of the diaphragm.
Stimulated tracheal pressure during electromagentical stimulation of the phrenic nerve | Study duration (10 days)
  Stimulated tracheal pressure is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Rapid Shallow Breathing Index (RSBI) record and evaluation. | Study duration (10 days)
  Progression of RSBI during 10 days after subject inclusion, based on the mechanical ventilation parameters (Tidal volume) and the ICU continuous monitoring system (Respiratory Rate).
Lung compliance during electromagentical stimulation of the phrenic nerve | 10 days
  Lung compliance is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Lung resistance during electromagentical stimulation of the phrenic nerve | 10 days
  Lung resistance is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Maximal inspiratory pressure (MIP) during electromagnetical stimulation of the phrenic nerve. | Study duration (10 days)
  MIP is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
Expiratory and Inspiratory Diaphragm Thickness measured by Ultrasound | Study duration (10 days)
  Diaphragm Thickness measured by Ultrasound as a baseline parameter for muscle atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be requested on reasonable scientific request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of scientific manuscript.
Access Criteria: Deidentified data can be requested on reasonable scientific request.

REFERENCES:
- [Derived] Panelli A, Grimm AM, Krause S, Verfuss MA, Ulm B, Grunow JJ, Bartels HG, Carbon NM, Niederhauser T, Weber-Carstens S, Brochard L, Schaller SJ. Noninvasive Electromagnetic Phrenic Nerve Stimulation in Critically Ill Patients: A Feasibility Study. Chest. 2024 Sep;166(3):502-510. doi: 10.1016/j.chest.2024.02.035. Epub 2024 Feb 24. PMID 38403186